CLINICAL TRIAL: NCT00184899
Title: The Potential Role for Adenosine in the Haemodynamic Effects of Free Fatty Acids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: Intralipid-Ado; ZonMw Nr. 920-03-249
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2007-03-01 (Estimated); Status verified 2007-02

CONDITIONS: Obesity; Metabolic Syndrome X
Keywords: free fatty acids; vasodilation; sympathetic activity
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Aneurysm | interventions — Heparin

INTERVENTIONS:
Drug: Intravenous infusion of Intralipid/heparin
Drug: Intravenous infusion of Glycerol/heparin

SUMMARY:
The metabolic syndrome is associated with hyperdynamic circulation and sympathetic activation. Recently, Bakker et al. (Atherosclerosis 2002) described the hypothesis that free fatty acids are responsible for this association. The investigators hypothesize that in patients with obesity and the metabolic syndrome, an increased intracellular concentration of long-chain fatty acyl (LCFA)-CoA (the intracellular equivalent of free fatty acids) induces an increase in adenosine. Adenosine receptor stimulation, in turn, induces vasodilation and sympathetic activation.

The investigators aimed to assess this effect of free fatty acids on the adenosine system in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Pregnancy
* Asthma
* Use of medication
* Cardiovascular/pulmonary disease and diabetes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-08; Study Completion 2006-08

PRIMARY OUTCOMES:
Forearm blood flow
Vasoactive effect of caffeine
Sympathetic activity (noradrenaline spillover, spectral analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Smits, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Background] Bakker SJ, Gans RO, ter Maaten JC, Teerlink T, Westerhoff HV, Heine RJ. The potential role of adenosine in the pathophysiology of the insulin resistance syndrome. Atherosclerosis. 2001 Apr;155(2):283-90. doi: 10.1016/s0021-9150(00)00745-0. PMID 11254897